CLINICAL TRIAL: NCT06879457
Title: Empowering Homebound Older Adults in Self-care Using a Mobile Health-assisted, Person-centred Care Approach: A Hybrid Effectiveness-implementation Design
Brief Title: mHealth Person-centred Self-care Support for Homebound Older Adults: A Hybrid Effectiveness-implementation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20240718004
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mobile Health; Person-Centred Care; Self-Care; Homebound; Older Adults

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group emphasizes shared decision-making, goal-setting, and interdisciplinary support. The NCM will co-develop self-care plans with participants.
  Interventions: Behavioral: PCC-based mHealth-assisted self-care support intervention
- Control Group (Active Comparator): The control group does not include shared decision-making or personalized goal-setting. Self-care plans will be developed solely by the nurse case manager (NCM).
  Interventions: Behavioral: Provider-led mHealth-assisted self-care support intervention

INTERVENTIONS:
Behavioral: PCC-based mHealth-assisted self-care support intervention — Participants receive six bi-weekly WhatsApp video call sessions with a NCM over three months, using a person-centred care (PCC) approach.
  Arms: Intervention Group
Behavioral: Provider-led mHealth-assisted self-care support intervention — Participants receive six bi-weekly WhatsApp video call sessions with a NCM over three months, based on the conventional provider-led model.
  Arms: Control Group

SUMMARY:
The aim of the study is to evaluate the effectiveness and implementation of the mobile health (mHealth)-assisted, person-centred care (PCC) self-care support programme for homebound older adults. The researcher will compare PCC approach to a conventional care provider-led model. Participants (n = 130) will receive the intervention of six bi-weekly WhatsApp video call sessions over three months with nurse case managers (NCMs).

DETAILED DESCRIPTION:
This hybrid effectiveness-implementation, cluster-randomized controlled trial evaluates a mHealth-assisted, PCC self-care support programme for homebound older adults in Hong Kong. Participants (n = 130) receive six bi-weekly WhatsApp video call sessions with NCMs over three months. The study compares a PCC-based approach with a conventional provider-led model. Effectiveness outcomes include self-efficacy, functional independence, and psychosocial well-being. Implementation is assessed using the RE-AIM framework. Findings will inform scalable, digital health interventions for aging populations, improving functional independence, self-care engagement, and healthcare accessibility for homebound older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older;
* Unable to leave home more than twice per week due to physical or functional health problems;
* Own and have basic proficiency in using a smartphone;
* Speak Cantonese;
* Indicate sufficient cognitive ability; and
* Be moderately frail or below.

Exclusion Criteria:

* Unable to hear, see, or communicate effectively;
* Be completely bed-bound; or
* Reside in an area without stable internet coverage.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-efficacy assessed using the Chinese version of the General Self-Efficacy Scale | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean score on self-efficacy.
Change in instrumental activities of daily living assessed using the Chinese version of the Lawton Instrumental Activities of Daily Living Scale | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean score on instrumental activities of daily living.

SECONDARY OUTCOMES:
Change in quality of life assessed using the Chinese version of the 12-item Short Form Health Survey version 2 | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean score on quality of life.
Change in psychological distress assessed using the Chinese version of 21-item Depression Anxiety Stress Scale | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean score on psychological distress.
Change in perceived loneliness assessed using the Chinese version of the UCLA 3-item Loneliness Scale | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean score on perceived loneliness.
Change in functional mobility assessed using the Timed Up and Go Test | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Time in seconds.
Change in sedentary behaviour assessed using the Chinese version of the Sedentary Behaviour Questionnaire for Elderly | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Mean hours per day.
Change in frequency of healthcare utilization assessed using the self-reported healthcare utilization survey | At baseline, 3 months post-intervention , and 6 months post-intervention.
  Unit of Measure: Number of visits.
Participant reach and recruitment success measured by recruitment records | At baseline.
  Unit of Measure: Percentage of eligible enrollment.
Participant satisfaction with the intervention assessed using the Chinese version of four-dimension Client Satisfaction Questionnaire | At 3 months post-intervention and 6 months post-intervention.
  Unit of Measure: Mean score on satisfaction.
Service provider acceptability and adoption of person-centred care approach measured by focus group interview | At 3 months post-intervention.
  Unit of Measure: Thematic analysis of interview records.
Implementation fidelity and adherence to person-centred care principles measured by session recordings and fidelity checklist | Ongoing monitoring during intervention.
  Unit of Measure: 1). Number and reasons for missed sessions; 2). Percentage of sessions meeting fidelity criteria.
Long-term maintenance and retention of participants measured by cost-effectiveness analysis and retention and dropout records | At 6 months post-intervention.
  Unit of Measure: 1). Incremental cost-effectiveness ratio (ICER) per additional quality adjusted life year (QALY) gained; 2). Number and reasons of dropout.
Barriers and Facilitators to the intervention measured by focus group interview | At 3 months post-intervention.
  Unit of Measure: Thematic analysis of interview records.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Arkers Wong, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- Yan Oi Tong, Hong Kong, Hong Kong